CLINICAL TRIAL: NCT05110963
Title: Intervention to Improve HIV Care Retention and Antiretroviral Adherence in Stigmatized Environments
Brief Title: Intervention to Improve HIV Care Retention by Addressing Stigma Stigmatized Environments
Acronym: Yomelela
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H19-157
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: HIV I Infection
Keywords: HIV

STUDY DESIGN:
Intervention Model Description: Behavioral skills training to improve medication adherence
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study condition masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Uniform Standard of Care Counseling (Placebo Comparator): Routine HIV counseling services available to patients with protocol delivered services. Three sessions of patient education monitored for protocol adherence.
  Interventions: Behavioral: Uniform Standard of Care Counseling
- Behavioral Self-Regulation Skills Counseling (Active Comparator): Mobile phone-delivered counseling grounded in Behavioral Self- Regulation Theory to improve retention in HIV care and HIV viral suppression. Counseling is delivered by lay counselors in differentiated health care context. This is a culturally tailored adaptation of CDC disseminated Phone-Delivered Support Counseling for HIV treatment Adherence.
  Interventions: Behavioral: Behavioral Self-Regulation Skills Counseling
- Behavioral Self-Regulation Skills Counseling + Stigma Management (Experimental): Mobile phone-delivered counseling grounded in Behavioral Self- Regulation Theory with stigma management to improve retention in HIV care and HIV viral suppression. Counseling is delivered by lay counselors in differentiated health care context with added components directly targeting stigma-related experiences and concerns.
  Interventions: Behavioral: Behavioral Self-Regulation Skills Counseling + Stigma Management

INTERVENTIONS:
Behavioral: Uniform Standard of Care Counseling — Routine HIV counseling services available to patients with protocol delivered services. Three sessions of patient education monitored for protocol adherence
  Arms: Uniform Standard of Care Counseling
Behavioral: Behavioral Self-Regulation Skills Counseling — Mobile phone-delivered counseling grounded in Behavioral Self- Regulation Theory to improve retention in HIV care and HIV viral suppression. Counseling is delivered by lay counselors in differentiated health care context. This is a culturally tailored adaptation of CDC disseminated Phone-Delivered Support Counseling for HIV treatment Adherence.
  Arms: Behavioral Self-Regulation Skills Counseling
Behavioral: Behavioral Self-Regulation Skills Counseling + Stigma Management — Mobile phone-delivered counseling grounded in Behavioral Self- Regulation Theory with stigma management to improve retention in HIV care and HIV viral suppression. Counseling is delivered by lay counselors in differentiated health care context with added components directly targeting stigma-related experiences and concerns.
  Arms: Behavioral Self-Regulation Skills Counseling + Stigma Management

SUMMARY:
Retention in care and persistent adherence to antiretroviral therapy are necessary for the successful treatment of HIV infection. HIV-related stigma is a known impediment to the care and health outcomes of people living with HIV. The proposed study will test theory-based interventions designed to manage HIV stigma in order to improve care retention and medication adherence in communities with high-levels of HIV-related stigma.

DETAILED DESCRIPTION:
This trial is conducting a randomized test of a behavioral self-management intervention designed to improve HIV treatment outcomes in people living with HIV in stigmatized contexts. The trial includes a control arm and a non-stigma enhanced treatment adherence intervention arm. Participants living in an economically under-resourced area of South Africa are recruited through clinical care settings. The goal of the research is to examine whether directly addressing HIV stigma and medication adherence management improves treatment outcomes beyond those observed from a standard behavioral intervention without added stigma-addressing components.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. current clinic visit to receive cART in differentiated care outside of an adherence club
3. unsuppressed HIV at the most recent clinical testing confirmed in run-in
4. access to a phone

Exclusion Criteria:

Not meeting inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3771 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Medical Records of Care Appointments | 12-months
  Medical records are retrospectively collected for all scheduled care visits and coded for whether the visits were attended.The records are exclusively from the clinic where patients are initially recruited and with patient permission. The data obtained are expressed as the ratio of the number of care appointments attended relative to the number scheduled.
Blood Plasma RNA | 12-months
  Collection of dried blood spots are tested for HIV RNA (viral load) using PCR tests with results expressed as the number of RNA copies per mL of blood plasma.

SECONDARY OUTCOMES:
Antiretroviral Medication Adherence | 12-months
  Monthly unannounced phone assessments are used to conduct pill counts of antiretroviral medications. The pill counts are used to calculate the proportion of pills taken relative to the number of pills prescribed over a 30 day period.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Connecticut, Storrs, Connecticut
  - University of Connecticut Field Site, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalichman SC, Mathews C, Banas E, Kalichman MO. Stigma management intervention to improve antiretroviral therapy adherence: Phase-I test of concept trial, Cape Town South Africa. Glob Public Health. 2019 Aug;14(8):1059-1074. doi: 10.1080/17441692.2018.1552307. Epub 2018 Nov 30. PMID 30500309